CLINICAL TRIAL: NCT03846895
Title: The Role of the Micro-ablative Fractional CO2 Laser in Postmenopausal Women With Overactive Bladder Syndrome.
Brief Title: Vaginal CO2 Laser in Postmenopausal Women With Overactive Bladder Syndrome (OAB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Themos Grigoriadis, Assistant Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 303/16-04-2018
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Overactive Bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Group (Experimental): Microablative Fractional CO2 laser therapy at monthly intervals.
  The laser parameters that will be used are the following:
  1. Power: 40 watts,
  2. Dwell time:1000μs,
  3. Spacing 1000 μm,
  4. Depth: SmartStak parameter 3
  5. D-pulse mode.
  Interventions: Device: Microablative Fractional CO2 laser
- Placebo Group (Placebo Comparator): Placebo CO2 laser therapies at monthly intervals.
  The laser parameters that will be used are the following:
  1. Power: 0.5 watts,
  2. Dwell time:1000μs,
  3. Spacing 1000 μm,
  4. Depth: SmartStak parameter 1,
  5. Smart-pulse mode.
  Interventions: Device: Microablative Fractional CO2 laser

INTERVENTIONS:
Device: Microablative Fractional CO2 laser — 3 therapies intravaginally administered will be applied at monthly intervals
  Other Names: SmartXide2 V2LR, Monalisa Touch, DEKA, Florence, Italy

SUMMARY:
This study evaluates the clinical efficacy and symptom relief of vaginal fractional CO2 laser treatment in post-menopausal women with Overactive Bladder syndrome(OAB). Post-menopausal women with OAB syndrome who receive β3 adrenergic receptors (mirabegron 50mg) treatment, will be randomized in two groups. Half participants will receive active CO2 laser therapy, while the other half will receive placebo CO2 laser therapy.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (≥ 12 months of amenorrhea or FSH ≥ 40 after hysterectomy with bilateral oophorectomy) who receive β3 adrenergic receptors (mirabegron 50 mg) treatment for OAB
* Overactive bladder syndrome (OAB)

  * ≥ 3 months symptoms of urgency, with or without urinary incontinence, and ≥ 8 micturitions / 24h
  * At least 3 episodes of urgent urination (3rd-4th grade) as recorded in the patient perception intensity of urgency scale (PPiUS) during a 3 day urination calendar , with or without urinary incontinence.

Exclusion Criteria:

* Participants with:

  * Pelvic Organ Prolapse (POP) > stage II of the pelvic organ prolapse quantitation system (POP-Q)
  * Post void residual volume > 200 ml (measured by ultrasound)
  * Use of moisturizers or lubricants the last month
  * Use of vaginal estrogen in the last 6 months
  * Use of drugs for urinary incontinence
  * Use of psychotropic drugs
  * Symptomatic urinary tract infection
  * Active genital infection
  * Kidney or liver disease
  * Abnormal cardiac conduction, rate or rythm disorders
  * Diabetic neuropathy
  * Myasthenia gravis
  * History of malignant disease
  * Previous radio-chemo therapy

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 50 (Actual)
Dates: Start 2018-05-12 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Overactive Bladder questionaire (OAB-q) | 24 months
  It consists of an 8 item symptom bother scale section and a 25 item health related quality of life scale section (HRQL). Scores of each domain of the 2 sections range from 0 to 100. Higher scores indicate higher impact of overactive bladder symptoms.
3 days voiding diary | 24 months
  Assesses bladder function (frequency of micturition, urgency and urinary incontinence)

SECONDARY OUTCOMES:
King's Health Questionnaire (KHQ) | 24 months
  It has 3 sections: 1) general health and overall health related to urinary symptoms with 2 questions, 2) incontinence impact, role limitations, physical limitations, social limitations, personal limitations, emotions, sleep and energy, and severity coping measures with 19 questions and 3) bother or impact of urinary symptoms with 11 questions. Scores of each domain of the 2 sections range from 0 to 100. Scores of the third section range from 0 to 3. Higher scores indicate higher impact of urinary incontinence.
Patients Global Impression of Improvement (PGI-I) | 24 months
  It is a single question with 7 possible answers. Patients will chose the answer that applies at their impression of improvement after the laser therapy
Urogenital Distress Inventory questionaire (UDI-6) | 24 months
  It is a 6 item questionaire evaluating symptom distress of urinary incontinence and its impact on daily life. Scores range from 0 to 100. Higher scores indicate higher impact of urinary incontinence.
Pelvic Floor Impact Questionnaire-short form 7 (PFIQ-7) | 24 months
  It is a 7 item questionaire evaluating how much bladder symptoms affect their activities, relationships, and feelings.

CONTACTS AND LOCATIONS:
Overall Officials: Themos Grigoriadis, Assistant Professor, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Urogynecological Unit of Alexandra Hospital, Athens, Greece

REFERENCES:
- [Derived] Kypriotis K, Prodromidou A, Athanasiou S, Zacharakis D, Kathopoulis N, Douligeris A, Athanasiou V, Michala L, Grigoriadis T. Is the Addition of CO2 Laser to beta3-Adrenoceptor Agonist Mirabegron Effective in the Management of Overactive Bladder? Results of a Randomized Controlled Trial. Medicina (Kaunas). 2025 Jun 30;61(7):1198. doi: 10.3390/medicina61071198. PMID 40731828